CLINICAL TRIAL: NCT05386940
Title: Protein Kinase N1 Level Predicts Acute Kidney Injury in Patients Undergoing Cardiac Surgery
Brief Title: Protein Kinase N1 Level in Patients Undergoing Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2017004
Record Dates: First submitted 2022-05-15; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-01

CONDITIONS: Acute Kidney Injury; Extracorporeal Circulation; Complications; Surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PKN1 Tertile 1
  Interventions: Other: PKN1 level
- PKN1 Tertile 2
  Interventions: Other: PKN1 level
- PKN1 Tertile 3
  Interventions: Other: PKN1 level

INTERVENTIONS:
Other: PKN1 level — different PKN1 level after on-pump cardiac surgery

SUMMARY:
Acute kidney injury (AKI) is one of the most frequent major complications in patients undergoing cardiac surgery. CSA-AKI is independently related to increased perioperative mortality, increased hospital and ICU length of stay as well as heath care expenditure. Identification of relevant biomarkers may lead to early diagnosis and improve patient outcomes and health care costs. The pathophysiology of CSA-AKI is complex and ischemia-reperfusion injury is one of the important factors. Recently, it has been shown that Protein kinase N1 (PKN1) is associated with ischemia-reperfusion injury. In this study, relationship between PKN1 with the risk of CSA-AKI was analyzed and the predictive value of elevated level of PKN1 for early prediction of CSA-AKI was further evaluated.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is one of the most frequent major complications in patients undergoing cardiac surgery. The incidence of cardiac surgery-associated AKI (CSA-AKI) varies from 5% to 42% and is the second leading cause of AKI (after sepsis) in the intensive care unit (ICU). CSA-AKI is independently related to increased perioperative mortality, increased hospital and ICU length of stay as well as heath care expenditure. Early detection of CSA-AKI could improve patient outcomes and health care costs through targeted interventions. Thus, identification of relevant biomarkers may lead to early diagnosis. The pathophysiology of CSA-AKI is complex and ischemia-reperfusion injury is one of the important factors. Recently, it has been shown that Protein kinase N1 (PKN1) is associated with ischemia-reperfusion injury. Nowadays, little is known about relationship between PKN1 and CSA-AKI. In this study, relationship between PKN1 with the risk of CSA-AKI was analyzed and the predictive value of elevated level of PKN1 for early prediction of CSA-AKI was further evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients (≥18 years old) underwent on-pump cardiac surgery
* admitted to ICU immediately after surgery

Exclusion Criteria:

* Patients younger than 18 years
* with prior AKI
* end-stage kidney disease
* need for chronic hemodialysis
* pregnant patients
* unable to give written consent for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (≥18 years old) underwent on-pump cardiac surgery and admitted to ICU immediately after surgery
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2021-03-14 (Actual); Study Completion 2021-03-14 (Actual)

PRIMARY OUTCOMES:
the development of CSA-AKI | 1 Week
  the development of CSA-AKI

SECONDARY OUTCOMES:
AKI severity | 1 Week
  AKI stage 1，stage 2，stage 3
need for RRT | 1 Week
  Reflect kidney function
duration of AKI (≥7 days) | 1 Week
  Reflect kidney function
length of ICU stay | up to 28 days
  Reflect patient prognosis
post-operative hospital stay | up to 28 days
  Reflect patient prognosis

CONTACTS AND LOCATIONS:
Overall Officials: ZhiYong Peng, Study Director — Department of Critical Care Medicine, Zhongnan Hospital of Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No